CLINICAL TRIAL: NCT03205670
Title: An Open Prospective Clinical Study on Safety and Efficacy of Surgical Treatment of Patients With Anterior Urethral Stricture Using a Tissue-engineered Construct Based on Autologous Buccal Mucosa Cells and Matrix From Reconstituted Collagen and Reinforcing Polylactoglycolide Fibers
Brief Title: Tissue-engineered Construct Based on Buccal Mucosa Cells and Matrix From Collagen and Polylactoglycolide Fibers
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Denis Butnaru, MD, Director, I.M. Sechenov First Moscow State Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SU-IRM-2017-0001
Record Dates: First submitted 2017-06-26; First posted 2017-07-02 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Urethral Stricture
Keywords: Autologous Cells; Buccal Mucosa; Urethroplasty; Tissue-engineered Construct; Hybrid matrix; Collagen; Polylactoglycolide Fibers
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Urethroplasty with a tissue-engineered construct (Experimental): The investigators will take a sample of the buccal mucosa to isolate epithelial cells. Autologous cells will be seeded on a hybrid matrix. Urethroplasty with this tissue-engineered construct will be performed. This is a single arm study with no control. All patients will undergo the surgical operation.
  Interventions: Procedure: Urethroplasty with a tissue-engineered construct

INTERVENTIONS:
Procedure: Urethroplasty with a tissue-engineered construct — The investigators will perform urethroplasty with the tissue-engineered construct - epithelial cells isolated from patient's buccal mucosa and seeded on a collagen-polylactoglycolide matrix.

SUMMARY:
This study investigates safety and efficacy of surgical treatment of patients with anterior urethral stricture using a tissue-engineered construct based on autologous buccal mucosa cells and matrix from reconstituted collagen and reinforcing polylactoglycolide fibers. This is a single arm study with no control. Success will be assessed via objective and subjective methods; complications will be tallied in a standardized fashion. Outcomes will be measured at five years.

DETAILED DESCRIPTION:
Treatment of urethral strictures longer than 2 cm is an actual clinical challenge. In this case, the common method is replacement surgery using a buccal mucosa graft. However, the main disadvantage of this method is associated with limited donor resources and donor site morbidity.

The aim of this study is to assess safety and efficacy of surgical treatment of patients with anterior urethral stricture using a tissue-engineered construct. The construct consists of autologous buccal mucosa cells and matrix from reconstituted collagen and reinforcing polylactoglycolide fibers. Patients will be followed up for 5 years within this study. The follow-up regimen includes retrograde and pericatheter urethrography, voiding cystourethrography, uroflowmetry, biopsy, and quality of life monitoring. Telephone follow-up will take place in between these assessments.

The data obtained from this study will have practical implications for the urethral stricture treatment and will be based on the principles of evidence-based medicine.

ELIGIBILITY:
Inclusion Criteria:

* Patient signed informed consent form
* Diagnosed anterior urethral stricture longer than 2.0 cm and shorter than 4.0 cm
* At least one prior internal optical urethrotomy and/or urethral bougienage

Non-inclusion Criteria:

* Acute infectious diseases
* Patient with decompensated heart and renal failure
* Patient with non-compensated diabetes mellitus
* Patient with malignant tumor
* Patient with polyvalent allergy
* Mental disorders
* Post traumatic urethral strictures
* Subtotal and total urethral strictures
* Sexually transmitted infections
* Hypersensitivity to any components of tissue-engineered constructs
* Any clinical state which does not ensure the safe implementation of study procedure (investigator's view)
* Other associated urethral strictures
* Laboratory markers of active urethritis

Exclusion Criteria:

* Patient's refusal from the further participation in trial
* Confirmed syphilis, HIV, hepatitis B or C infections
* Patient who cannot be regularly examined due to any circumstances

Ages: 18 Years to 78 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Serious adverse events | 4 weeks after surgery
  Frequency, type and severity of serious adverse events (SAE)
Serious adverse reactions | 4 weeks after surgery
  Frequency, type and severity of serious adverse reactions (SAR)

SECONDARY OUTCOMES:
Retrograde urethrography | 5 years
  Influence of the surgery on the urethral lumen
Voiding cystourethrography | 5 years
  Full assessment of the urethral lumen after the surgery
Pericatheter urethrography | 4 weeks after surgery
  Assessment of absence or presence of contrast medium leakage outside the urethra
Biopsy | 4 months after surgery
  Control of anatomical urethral structure in the intervention place
Urodynamic changes via uroflowmetry - 1 | 5 years
  Influence of the surgery on urinary flow rate: maximum flow rate
Urodynamic changes via uroflowmetry - 2 | 5 years
  Influence of the surgery on urinary flow rate: average flow rate
Urodynamic changes via uroflowmetry - 3 | 5 years
  Influence of the surgery on urinary flow rate: total volume voided
Urodynamic changes via uroflowmetry - 4 | 5 years
  Influence of the surgery on urinary flow rate: maximum flow time
Quality of life monitoring - 1 | 5 years
  Quality of life estimated by validated questionnaires: Short Form (SF-36)
Quality of life monitoring - 2 | 5 years
  Quality of life estimated by validated questionnaires: International Prostatic Symptom Score (IPSS)

CONTACTS AND LOCATIONS:
Overall Officials: Denis Butnaru, Dr., Principal Investigator — Sechenov First Moscow State Medical University; Andrey Vinarov, Dr., Prof., Principal Investigator — Sechenov First Moscow State Medical University
Locations (1):
- Sechenov University, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided